CLINICAL TRIAL: NCT01553448
Title: The Role of Stroma-Derived Soluble TßRIII in Neuroblastoma
Brief Title: Studying Gene Expression in Samples From Younger Patients With Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL12B6; COG-ANBL12B6 (Other: Children's Oncology Group); CDR0000728527 (Other: Clinical Trials.gov); ANBL12B6 (Other: Children's Oncology Group); NCI-2012-00706 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-03-13; First posted 2012-03-14 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Neoplastic Syndrome; Neuroblastoma
Keywords: disseminated neuroblastoma; hereditary neuroblastoma; localized resectable neuroblastoma; localized unresectable neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neoplasms; Neuroblastoma | interventions — Gene Expression Profiling; Enzyme-Linked Immunosorbent Assay; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: enzyme-linked immunosorbent assay
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

PURPOSE: This research trial studies gene expression in samples from younger patients with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether TβRIII expression and TGF-β signaling decrease in advanced-stage neuroblastoma (NBL) and whether these changes are confined to the Schwannian stroma.
* Determine whether sTβRIII levels and TGF-β signaling correlate with NBL stage, tumor stroma content, surface TβRIII expression, and TGF-β signaling.

OUTLINE: Archived paraffin-embedded tissue and plasma samples are analyzed for TβRIII expression, TGF-β signaling, and SMAD3 expression and phosphorylation by immunohistochemistry, enzyme-linked immunosorbent assay (ELISA), and other assays. Surface expression of TβRIII in the neuroblastic and stromal tumor components are correlated with matched circulating levels of soluble TβRIII. Results are then correlated with each patient's outcome data, including stage.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tissue samples and matched plasma samples available from 1 of the following groups:

  * Patients with low-stage (International Neuroblastoma Staging System [INSS] stage 1 or 2) neuroblastoma (NBL)
  * Patients with advanced-stage (INSS stage 3 or 4) NBL
  * Patients with stage 4S NBL
* Clinical and/or outcome data associated with the tissue and plasma samples including INSS stage, age, MYCN amplification status, chromosomal alterations, and 5-year survival, if known

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with low-stage (International Neuroblastoma Staging System [INSS] stage 1 or 2) neuroblastoma (NBL), patients with advanced-stage (INSS stage 3 or 4) NBL, or patients with stage 4S NBL
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Expression of TβRIII in the neuroblastic tumor and stroma of patients with advanced-stage NBL
Correlation between TβRIII levels and TGF-β signaling correlate with NBL stage, tumor stroma content, surface TβRIII expression, and TGF-β signaling

CONTACTS AND LOCATIONS:
Overall Officials: Gerard C. Blobe, MD, PhD, Principal Investigator — Duke University